CLINICAL TRIAL: NCT02054468
Title: Rocuronium Dose Finding Study After Single-shot or Steady-state Propofol
Brief Title: Rocuronium Dose Finding Study After Single-shot or Steady-state Propofol Anesthesia
Acronym: ROSANNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSANNA
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Neuromuscular Blockade; Anesthesia
Keywords: Muscle relaxant, Rocuronium, TIVA, Propofol
MeSH Terms: conditions — Muscle Hypotonia | interventions — Propofol; Remifentanil; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-shot-Propofol & Remifentanil (Active Comparator): Induction group: A single-shot propofol induction dose with remifentanil infusion followed by injection of rocuronium (for doses, please see interventions). Airway: tracheal intubation
  Interventions: Drug: Single-Shot Propofol; Drug: Remifentanil infusion; Drug: Rocuronium (0.07mg/kg/body mass); Drug: Rocuronium (0.1mg/kg/body mass); Drug: Rocuronium (0.15mg/kg/body mass); Drug: Rocuronium (0.2mg/kg/body mass); Drug: Rocuronium (0.3mg/kg/body mass); Drug: Rocuronium (0.45mg/kg/body mass)
- 30min infusion Propofol & Remifentanil (Experimental): Maintenance group: 30min of total intravenous anesthesia (TIVA) with propofol and remifentanil before rocuronium (for doses, please see interventions) is administered. Airway: tracheal intubation/laryngeal mask
  Interventions: Drug: 30min infusion Propofol; Drug: Remifentanil infusion; Drug: Rocuronium (0.07mg/kg/body mass); Drug: Rocuronium (0.1mg/kg/body mass); Drug: Rocuronium (0.15mg/kg/body mass); Drug: Rocuronium (0.2mg/kg/body mass); Drug: Rocuronium (0.3mg/kg/body mass); Drug: Rocuronium (0.45mg/kg/body mass)

INTERVENTIONS:
Drug: Single-Shot Propofol — Single-shot propofol induction dose (1.5-2.5mg/kg body mass)
  Other Names: 2,6-Diisopropylphenol
  Arms: Single-shot-Propofol & Remifentanil
Drug: 30min infusion Propofol — 30min of propofol infusion (4-6mg/kg/h)
  Other Names: 2,6-Diisopropylphenol
  Arms: 30min infusion Propofol & Remifentanil
Drug: Remifentanil infusion — Remifentanil infusion (0.1-0.2µg/kg/min)
  Other Names: Ultiva®
Drug: Rocuronium (0.07mg/kg/body mass) — Rocuronium (0.07mg/kg/body mass)
  Other Names: Esmeron
Drug: Rocuronium (0.1mg/kg/body mass) — Rocuronium (0.1mg/kg/body mass)
  Other Names: Esmeron
Drug: Rocuronium (0.15mg/kg/body mass) — Rocuronium (0.15mg/kg/body mass)
  Other Names: Esmeron
Drug: Rocuronium (0.2mg/kg/body mass) — Rocuronium (0.2mg/kg/body mass)
  Other Names: Esmeron
Drug: Rocuronium (0.3mg/kg/body mass) — Rocuronium (0.3mg/kg/body mass)
  Other Names: Esmeron
Drug: Rocuronium (0.45mg/kg/body mass) — Rocuronium (0.45mg/kg/body mass)
  Other Names: Esmeron

SUMMARY:
This study is designed to determine the effective-doses ED-50 and ED-95 (the doses required for a 50% and 95% twitch inhibition, respectively) of the non-depolarizing muscle relaxant rocuronium after single-shot or steady-state propofol anesthesia in a clinical setting.

DETAILED DESCRIPTION:
Neuromuscular blocking agents are worldwide used as a standard component of a modern balanced anesthesia regime. They are administered to facilitate tracheal intubation, reduce laryngeal trauma and optimize surgical conditions. The dose usually recommended to facilitate tracheal intubation approximates at least two times the drug´s effective dose ED-95 (the dose required for a 95% effect) depending on the choice of the neuromuscular blocking agent. This overdose is administered to induce a very deep paralysis with a fast onset of action providing clinically acceptable intubating conditions. Moreover, our clinical experience has shown that the dose-relationship of a neuromuscular blocking agents estimated during steady-state anesthesia does not necessarily correlate with the dose-response curve of the same drug during anesthetic induction. Therefore, a discrepancy between the applied dose and the clinical outcome measure, the intubating conditions, becomes apparent. This might be related to effects of the co-administered anesthetics at the neuromuscular junction. While inhaled anesthetics augment the paralyzing effects of non-depolarizering muscle relaxants in a dose-dependent fashion and depend on the duration of anesthesia, little is known about the interactions of the intravenous anesthetic propofol with the non-depolarizing blocking agent rocuronium. We hypothesize that the intravenous administration of propofol also influences the potency of rocuronium dependant on the duration of its application.

This study, therefore, is designed to determine the dose-response relationship of rocuronium after single-shot or steady-state propofol anesthesia in a clinical setting. The primary endpoints are the ED-50s and ED-95s of rocuronium during anesthetic induction with a single-shot propofol and after 30minutes of steady-state propofol anesthesia. The secondary endpoints are the slopes and the intercepts of the respective dose-response-curves, the onset and duration of muscle paralysis and the recovery from neuromuscular blockade.

Materials & Methods

We will investigate patients scheduled for elective low-risk surgical procedures under general anesthesia. Patients will be allocated to two experimental groups. After neuromuscular monitoring is established under remifentanil infusion, patients of the group "Induction" will receive a single-shot propofol followed by injection of rocuronium and endotracheal intubation. Patients of the group "Maintenance" will be anaesthetized with an induction dose of propofol followed by 30 minutes of total intravenous anesthesia (TIVA: propofol/ remifentanil) before rocuronium is administered. Airway will be managed using a laryngeal mask or tracheal intubation.

During surgery, anesthesia will be maintained with TIVA. Onset and duration of neuromuscular blockade and spontaneous recovery will be monitored with electromyography.

Postoperatively, patients will be monitored for 60 minutes in our post-anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for a low risk-surgical procedure under general anesthesia
2. Patients ASA physical status I-III
3. Patients older than 18years
4. Patients having given informed consent to the study

Exclusion Criteria:

1. Patients who decline to give informed consent to the study
2. Known or suspected allergy towards anesthetics or rocuronium
3. Pregnant and breastfeeding women
4. Known or suspected neuromuscular disease
5. Burn injury prior to the investigation
6. Anatomic and functional malformations with expected difficult intubation
7. Anorexia, Bulimia nervosa, Malnutrition
8. Heart failure
9. Use of drugs that interfere with muscle relaxant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
ED-50 of rocuronium | Anesthesia time during their surgical procedure (=arrival in the OR until discharge from the post-anesthesia care unit), ca. 180min
  The primary outcome measure is the 1) ED-50 of rocuronium during anesthesia induction with propofol and after steady-state propofol anesthesia
ED-95 of rocuronium | Anesthesia time during their surgical procedure (=arrival in the OR until discharge from the post-anesthesia care unit), ca. 180min
  The primary outcome measure is 2) the ED-95 of rocuronium during anesthesia induction with propofol and after steady-state propofol anesthesia

SECONDARY OUTCOMES:
Pharmacodynamics of rocuronium (composite outcome measure) | Anesthesia time during their surgical procedure (=arrival in the OR until discharge from the post-anesthesia care unit), ca. 180min
  The secondary outcome measures are the slopes and the intercepts of the dose-response-curves for rocuronium, the onset and duration of muscle paralysis and the recovery from neuromuscular blockade.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, M.D., Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München, Germany
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Naguib M, Seraj M, Abdulrazik E. Pipecuronium-induced neuromuscular blockade during nitrous oxide-fentanyl, enflurane, isoflurane, and halothane anesthesia in surgical patients. Anesth Analg. 1992 Aug;75(2):193-7. doi: 10.1213/00000539-199208000-00007. PMID 1321569
- [Background] Viby-Mogensen J, Jorgensen BC, Ording H. Residual curarization in the recovery room. Anesthesiology. 1979 Jun;50(6):539-41. doi: 10.1097/00000542-197906000-00014. No abstract available. PMID 156513
- [Background] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Background] Eikermann M, Blobner M, Groeben H, Rex C, Grote T, Neuhauser M, Beiderlinden M, Peters J. Postoperative upper airway obstruction after recovery of the train of four ratio of the adductor pollicis muscle from neuromuscular blockade. Anesth Analg. 2006 Mar;102(3):937-42. doi: 10.1213/01.ane.0000195233.80166.14. PMID 16492855
- [Background] Hemmerling TM, Le N, Decarie P, Cousineau J, Bracco D. Total intravenous anesthesia with propofol augments the potency of mivacurium. Can J Anaesth. 2008 Jun;55(6):351-7. doi: 10.1007/BF03021490. PMID 18566198
- [Background] Robertson EN, Fragen RJ, Booij LH, van Egmond J, Crul JF. Some effects of diisopropyl phenol (ICI 35 868) on the pharmacodynamics of atracurium and vecuronium in anaesthetized man. Br J Anaesth. 1983 Aug;55(8):723-8. doi: 10.1093/bja/55.8.723. PMID 6136286